CLINICAL TRIAL: NCT05909319
Title: Identification and Verification of Neutrophil Extracellular Trap Net Related Markers in Acute-on-chronic Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-3-14 version V1.0
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-04

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Neutrophil extracellular traps
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACLF

SUMMARY:
Acute-on-chronic liver failure (ACLF) refers to the acute deterioration of liver function in patients with chronic liver disease. Neutrophils are a major component of the innate immune system, and previous studies have revealed enhanced production of neutrophil extracellular traps (NETs) in ACLF. However, there is still a lack of systematic research on the correlation between NETs and the prognosis of ACLF. We screened NETs related biomarkers through bioinformatics analysis, which play an important role in the diagnosis of ACLF. This study will explore whether these NETs related biomarkers also play an important role in the prognosis of ACLF and further investigate their role in the pathogenesis of ACLF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria of Chinese Group on the Study of Severe Hepatitis B (COSSH) for acute-on-chronic liver failure

Exclusion Criteria:

1. Age greater than 75 years old
2. liver cancer
3. previous liver transplantation
4. other serious extrahepatic organ diseases
5. uncontrolled bacterial infections.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who meet the diagnostic criteria of Chinese Group on the Study of Severe Hepatitis B (COSSH) for acute-on-chronic liver failure
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-25 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days
  mortality of patients with ACLF
mortality | 90 days
  mortality of patients with ACLF
mortality | half a year
  mortality of patients with ACLF